CLINICAL TRIAL: NCT04600986
Title: The Effect of Repeated Doses of a GnRH Agonist on Oocyte Triggering in Antagonist Protocol for Patients With Polycystic Ovary Syndrome: a Randomized Clinical Trial)
Brief Title: Repeated Doses of GnRH Agonist as Oocyte Triggering in Antagonist Protocol for Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Female infertility (97000253)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New oocyte triggering (Experimental): The final oocyte maturation will be triggered with a single dose of 0.2 mg s.c triptorelin (decapeptyl) and in addition a repeat dose of 0.1 mg s.c triptorelin (decapeptyl) will prescribed 12 h following the first dose.
  Interventions: Other: Repeated dose of GnRH agonist
- Routine oocyte trigering (Other): The final oocyte maturation will be triggered with a single dose of 0.2 mg s.c triptorelin (decapeptyl), 35 h prior to oocyte retrieval.
  Interventions: Other: Repeated dose of GnRH agonist

INTERVENTIONS:
Other: Repeated dose of GnRH agonist — 0.2 mg triptorelin plus a repeat dose of 0.1 mg 12 hours following the first dose.

SUMMARY:
This is a prospective, randomized, proof-of-concept study, designed to compare the IVF results in patients diagnosed with polycystic ovarian syndrome (PCOS) defined as per the ESHRE/ASRM Rotterdam criteria (2003) undergoing in-vitro fertilization/ intracytoplasmic sperm injection (IVF/ICSI) in antagonist protocol. Patients were randomized into two groups. Group A: single dose of GnRHa 0.2 mg, 35 h prior to oocyte retrieval, and Group B: 0.2 mg GnRHa 35 h prior to oocyte retrieval + a repeat dose of 0.1 mg 12 h following the 1st dose. 12 h post-trigger, luteinizing hormone (LH), progesterone (P4) values will be estimated.

DETAILED DESCRIPTION:
The aim of this study was to establish if a second dose of GnRHa repeated 12 h following the initial dose optimizes the cycle outcome in terms of oocyte maturity in women with PCOS of Asian origin.

The study was approved by the institutional review board and written, informed consent will be obtained from each participant. Infertile women with a diagnosis of PCOS, who undergo the IVF / ICSI cycle are assigned to two groups randomly. The random method is that the statistician will be provided a blocked randomization list for the number of patients,and whenever an eligible patient is referred, a sealed envelope will be delivered to the clinical physician. The random allocation is concealed from the physician performing the IVF/ICSI treatment cycle. All patients will receive antagonist controlled ovarian stimulation protocol with same starting dose of gonadotropin. On the day of trigger, serum E2, LH, and P4 concentrations will be measured. When three lead follicles achieved 17-mm diameter, in group A, the final oocyte maturation will be triggered with a single dose of 0.2 mg s.c triptorelin (decapeptyl), 35 h prior to oocyte retrieval in both the groups and in Group B, a repeat dose of 0.1 mg 12 h following the first dose. Post-trigger, LH, and progesterone levels will be measured 12 h following the first dose of GnRHa and ovum-pick up day. Transvaginal ultrasound-guided oocyte pickup (OPU) will be performed 35 h following the first dose under intravenous sedation with single-lumen oocyte retrieval needle. Post pickup on days 4 and 7, an assessment for symptoms and signs of OHSS and patients will be advised to present at any time within 2 weeks of GnRHa administration.

In all subjects, IVF or ICSI will be performed according to the standard operating procedure. The fertilization will be assessed 18 h following ICSI or IVF by the appearance of two pronuclei. All embryos will be cryopreserved by vitrification in the form of blastocyst. The frozen embryo transfer (FET) cycles will be performed following pretreatment with oral contraceptive pills in an artificial cycle with a daily dose of orally administered 6 mg of estradiol. When the endometrium evaluated by TVS was >8 mm with triple-layer morphology, it is considered mature. This will be followed by endometrial priming with 5 days of injectable progesterone for blastocysts. The transfer will be performed using Sure-Pro Ultra catheter. Luteal-phase supplementation will be continued with vaginal progesterone and estradiol for 14 days and when pregnancy will be achieved till 10 weeks of gestation..

The primary outcome will be the maturity rate of the oocytes (the ratio of MII oocytes to the total number of oocytes retrieved) and oocyte yield. The secondary outcomes are fertilization rate, number and quality of blastocyst embryos, OHSS occurrence, and post-trigger serum LH (IU/L), and P4 (ng/mL) levels. In addition, implantation and clinical pregnancy rates will be also evaluated. Data collection will be performed by using questionnaires to be filled as per the available records and laboratory results. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS software version 20 for windows.

ELIGIBILITY:
Inclusion Criteria:

All PCOS patients defined as per the ESHE/ASRM Rotterdam criteria undergoing ovarian stimulation for IVF/ICSI using GnRH antagonist protocol:

1. Anticipated high ovarian response (serum E2> 3000 on trigger day)
2. Body mass index (BMI) >18 and <35 kg/m2
3. Willingness to participate in the study

Exclusion Criteria:

1. Severe male factor infertility
2. Patients with severe endometriosis
3. Donor cycles
4. Indication for preimplantation genetic diagnosis
5. Uterine abnormality or existing myoma greater than 5cm
6. couple's drug addiction

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Oocyte maturity rate | 24 hours post oocyte retrieval day
  Oocyte maturity was defined as the ratio of metaphase II (MII) oocytes to the number of collected oocytes in the patients undergoing with ICSI.
Oocyte yield | 34 to 36 hours post the first trigger with GnRHa
  Oocyte yield was defined as the ratio of the total number of collected oocytes to the number of follicles measuring ≥10 mm on the day of oocyte retrieval.

SECONDARY OUTCOMES:
Fertilization rate | 48 hours post IVF/ICSI
  Fertilization rate was defined as the ratio of normal fertilized oocytes (2PNs) to the number of oocytes used for fertilization.
Number and grading of blastocysts | 1 week after oocyte retrieval
  The number and grading of blastocysts suitable for biopsy and freezing
Post-trigger serum luteinizing hormone (LH) | 12 hours post trigger with the first injection of GnRHa
  Serum LH level 12 hours post first injection of GnRHa
Post-trigger serum progesterone (P4) | 12 hours post trigger with the first injection of GnRHa
  Serum P4 level 12 hours post first injection of GnRHa
Implantation rate | 1 month post embryo transfer
  The number of gestational sacs observed at trans-vaginal ultrasonography screening at 6 weeks of pregnancy divided by the number of embryos transferred.
Clinical pregnancy rate | 6-8 weeks of gestation
  Clinical pregnancy rate per transfer as defined by the presence of a gestational sac with heart beat on ultrasound at 6-8 weeks of gestation.
OHSS occurrence | 16 days post triggering
  Occurrence of ovarian hyperstimulation syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Hafezi, MD., Study Director — Department of Endocrinology and Female Infertility, Royan Institute; Hoora Hashemi, MD., Principal Investigator — Department of Endocrinology and Female Infertility, Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashemi SH, Hafezi M, Arabipoor A, Zareei M, Vesali S, Eftekhari-Yazdi P. Can We Harvest More Mature Oocytes by Repeating Gonadotropin-Releasing Hormone Agonist Doses in Polycystic Ovarian Syndrome Patients at Risk of OHSS in Antagonist Cycles? A Randomised Clinical Trial. Int J Fertil Steril. 2024 Jul 13;18(Suppl 1):48-54. doi: 10.22074/ijfs.2023.2008905.1513. PMID 39033370